CLINICAL TRIAL: NCT00328016
Title: Respiratory Adaptations to Behavioral Interventions in Elevated Blood Pressure
Brief Title: Breathe: Slow Paced Breathing to Lower Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0067
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2016-12

CONDITIONS: High Blood Pressure
Keywords: hypertension; high blood pressure; meditation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device Guided Breathing (Experimental): Individual breathing rate was determined from an expandable band around the torso connected to a commercially available device (RESPeRATE, Lod, Israel) that presented distinctive tones via earphones.
  Interventions: Device: RESPeRATE
- Control Group (Placebo Comparator): Control group were instructed to sit in the same manner passively attend to their breathing, and silently repeat 'one' during each exhalation. If other thoughts came to mind, they were instructed to calmly attend to their breathing.
  Interventions: Behavioral: Guided Breathing

INTERVENTIONS:
Behavioral: Guided Breathing — The participant will engage in daily 15 min sessions of meditative relaxation that involves quiet attention to breathing pattern with no attempt to manipulate breathing pattern
  Arms: Control Group
Device: RESPeRATE — The participant will be trained to perform a guided breathing task that involves a chest expansion sensor, battery-powered microcomputer, and earphones
  Arms: Device Guided Breathing

SUMMARY:
The purpose of this study is to investigate the nature of the physiological reasons for the decreases in resting blood pressure that can result from systematic practice of computer-guided breathing exercises or meditative relaxation.

DETAILED DESCRIPTION:
In this randomized clinical trial, persons with moderately elevated blood pressure were trained in either computer-guided breathing exercises or meditative relaxation to breathing. The computer-guided breathing exercise involves listening to tones of ascending and descending pitch to which breathing is entrained to low frequencies over a 15 minute interval. The meditative relaxation involves passive attention to natural breathing for the same duration. Participants will perform these breathing exercises daily at home for four weeks. Before and after the intervention, respiratory, cardiovascular, and urinary endogenous digitalis-like factors will be systematically recorded to determine the extent to which chronic neuroendocrine changes underlie the reductions in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Over 21 years
* Systolic blood pressure 130-160 or diastolic blood pressure 85-100

Exclusion Criteria:

* More than one antihypertensive medication
* Beta blockers, angiotensin converting enzyme inhibitors or angiotensin receptor blockers
* History of coronary artery disease, heart failure, stroke, angina or coronary revascularization
* Kidney disease, defined as plasma creatinine > 1.5mg/dL
* Diabetes, defined by insulin or oral hypoglycemic medication or blood sugar > 126mg/dL
* Pulmonary disease, defined as chronic obstructive pulmonary disease, bronchitis, asthma, or use of inhaler
* Upper respiratory infection during past 30 days
* Medication that affects central nervous system function
* Steroid use
* Current pregnancy or lactation within past six months
* Current birth control medication or hormone replacement therapy
* Condition that in the judgment of the Principal Investigator is incompatible with the research study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B. Ershler, M.D., Principal Investigator — NIA, Clinical research Unit
Locations (1):
- NIA Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual level data.

REFERENCES:
- [Background] Meles E, Giannattasio C, Failla M, Gentile G, Capra A, Mancia G. Nonpharmacologic treatment of hypertension by respiratory exercise in the home setting. Am J Hypertens. 2004 Apr;17(4):370-4. doi: 10.1016/j.amjhyper.2003.12.009. PMID 15062893
- [Background] Elliot WJ, Izzo JL Jr, White WB, Rosing DR, Snyder CS, Alter A, Gavish B, Black HR. Graded blood pressure reduction in hypertensive outpatients associated with use of a device to assist with slow breathing. J Clin Hypertens (Greenwich). 2004 Oct;6(10):553-9; quiz 560-1. doi: 10.1111/j.1524-6175.2004.03553.x. PMID 15470284
- [Background] Grossman E, Grossman A, Schein MH, Zimlichman R, Gavish B. Breathing-control lowers blood pressure. J Hum Hypertens. 2001 Apr;15(4):263-9. doi: 10.1038/sj.jhh.1001147. PMID 11319675
- [Background] Benson H. The Relaxation Response. New York: Avon Books, 1975
- [Result] Anderson DE, McNeely JD, Chesney MA, Windham BG. Breathing variability at rest is positively associated with 24-h blood pressure level. Am J Hypertens. 2008 Dec;21(12):1324-9. doi: 10.1038/ajh.2008.292. Epub 2008 Sep 25. PMID 18820654
- [Derived] Anderson DE, McNeely JD, Windham BG. Regular slow-breathing exercise effects on blood pressure and breathing patterns at rest. J Hum Hypertens. 2010 Dec;24(12):807-13. doi: 10.1038/jhh.2010.18. Epub 2010 Mar 4. PMID 20200548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 102 Subjects responded to advertising and were assessed for eligibility. Forty-four were enrolled and randomized. 23 were randomized to guided breathing and 21 were on the Control arm.
Groups:
- Device Guided Breathing: The Device Guided Breathing (DGB) group were instructed to sit comfortably with eyes closed and arms and legs uncrossed. Individual breathing rate was initially determined from an expandable band around the torso connected to a commercially available device (RESPeRATE, Lod, Israel) that presented distinctive tones via earphone. Each subject was instructed to inspire during ascending tones and expire during descending tones, following two training sessions, respiration, blood pressure and breathing parameters were monitored during a 10 min rest period, a 15 min guided breathing task period, and a 10 min recovery period.
- Control Group: The Control Group were instructed to sit in the same matter, passively attend to their breathing, and silently repeat 'one' during each exhalation. If thoughts came to mind, they were instructed to calmly refocus attention on breathing. Following two sessions of practice of passive attention to breathing, blood pressure and breathing parameters of each subject were also monitored during a 10 min baseline, 15 min passive attention to breathing and 10 min recovery period.
Period: Overall Study
Arm/Group | Device Guided Breathing | Control Group
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 44 subjects randomly assigned to treatment and control group, 12 subjects were excluded from data analysis due to either non-compliance with the intervention or abnormal breathing pattern during baseline session.
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Guided Breathing | Control Group | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 43
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Twelve subjects were excluded from data analysis due to either non-compliance with the intervention or abnormal breathing pattern during baseline session.
  years
    number analyzed (Participants) | 16 | 16 | 32
    (all) | 51.9 (11.6) | 54.5 (8.0) | 53.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants] — Population: Of the 44 subjects randomly assigned to treatment and control group, 12 subjects were excluded from data analysis due to either non-compliance with the intervention or abnormal breathing pattern during baseline session.
  participants
    United States: number analyzed (Participants) | 16 | 16 | 32
    United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Breathing Rate
Description: Breathing rate was monitored continuously via inductive plethysmography.
Time Frame: After 15 minutes of guided breathing or control task
Measure: Mean (Standard Error); unit: Breaths/minute
Groups:
- Device Guided Breathing: Practiced slow breathing using Guided Breathing Device
- Control Group: Practiced passive attention to breathing
Arm/Group | Device Guided Breathing | Control Group
Number analyzed (Participants) | 16 | 16
Breaths/minute | 9.4 (3.6) | 13.7 (4.7)

2. Secondary Outcome: Minute Ventilation
Description: Minute Ventilation was continuously monitored via inductive plethysmography
Time Frame: After 15 minutes of guided breathing or control task
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Device Guided Breathing | Control Group
Number analyzed (Participants) | 16 | 16
L/min | 7.6 (3.0) | 5.6 (1.8)

3. Secondary Outcome: End Tidal CO2 (PetCO2)
Description: End tidal CO2 was monitored continuously using a respiratory gas monitor
Time Frame: After 15 minutes of guided breathing or control task
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Device Guided Breathing | Control Group
Number analyzed (Participants) | 16 | 16
mmHg | 30.1 (5.6) | 36.5 (3.3)

ADVERSE EVENTS:
Groups:
- Device Guided Breathing: The Device Guided Breathing (DGB) group were instructed to sit comfortably with eyes closed and arms and legs uncrossed. Individual breathing rate was initially determined from an expandable band around the torso connected to a commercially available device (RESPeRATE, Lod, Israel) that presented distinctive tones via earphone. Each subject was instructed to inspire during ascending tones and expire during descending tones, following two training sessions, respiration, blood pressure and breathing parameters were monitored during a 10 min rest period, a 15 min guided breathing task period, and a 10 min recovery period during an experimental session on a subsequent day.
- Control Group: The Control Group were instructed to sit in the same matter, passively attend to their breathing, and silently repeat 'one' during each exhalation. If thoughts came to mind, they were instructed to calmly refocus attention on breathing. Following two sessions of practice of passive attention to breathing, blood pressure and breathing parameters of each subject were also monitored during a 10 min baseline, 15 min passive attention to breathing and 10 min recovery.
Arm/Group | Device Guided Breathing | Control Group
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes